CLINICAL TRIAL: NCT02079675
Title: Multi-center, Randomized, Double Blinded, Parallel Group, Placebo-controlled, Phase II Trial to Assess the Efficacy and Safety of SKI3246 in Subjects With Non-Constipation Irritable Bowel Syndrome
Brief Title: Study to Assess the Efficacy and Safety of SKI3246 in Subjects With Non-Constipation Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKI3246_IBS_II_2012
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Non-constipation Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SKI3246 Low Dose (Experimental): Intervention: Drug: SKI3246 Low Dose
  Interventions: Drug: SKI3246 Low Dose
- SKI3246 High Dose (Experimental): Intervention: Drug: SKI3246 High Dose
  Interventions: Drug: SKI3246 High Dose
- Placebo (Placebo Comparator): Intervention: Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKI3246 Low Dose — SKI3246 Low Dose will be taken for a 4-week duration (28 days) as 4 capsules a day: two capsules in the morning and two capsule in the evening
  Arms: SKI3246 Low Dose
Drug: SKI3246 High Dose — SKI3246 High Dose will be taken for a 4-week duration (28 days) as 4 capsules a day: two capsules in the morning and two capsule in the evening
  Arms: SKI3246 High Dose
Drug: Placebo — SKI3246 Placebo will be taken for a 4-week duration (28 days) as 4 capsules a day: two capsules in the morning and two capsule in the evening
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of different doses of SKI3246 compared with placebo in the treatment of patients with irritable bowel syndrome with non-constipation.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed as non-constipation by ROME III.
* Patients who voluntarily signed written informed consent may participate in the study.

Exclusion Criteria:

* Pregnant or lactating female.
* Patients with a history of inflammatory bowel disease.
* Severe neurological or psychological disease
* History of allergic reaction to the medications used in this study
* Use of other investigational drugs within 30 days prior to the study.
* Patients that investigators consider ineligible for this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Relief During the Double-Blind Treatment Phase Using the Subject Global Assessment (SGA) | 12 weeks

SECONDARY OUTCOMES:
Patient satisfaction using 5- Likert Scale | 4 weeks
Subject Self Reported Adequate Relief of Pain | 4 weeks
Mean Change From Baseline in Quality of Life as Measured by the Medical Outcomes Survey | 12 weeks
Visual Analog Scale (VAS) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jin Park, M.D., Study Chair — Gangnam Severance Hospital, Yonsei University College of Medicine
Locations (1):
- SK Chemicals, Seoul, South Korea